CLINICAL TRIAL: NCT01285271
Title: The Safety and Feasibility of Delivering Xenon to Patients Before and After Coronary Artery Bypass Graft Implantation: a Pilot Study
Brief Title: A Pre- and Post- Coronary Artery Bypass Graft Implantation Disposed Application of Xenon
Acronym: CArDiAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-017; 2010-023942-63 (EudraCT Number)
Record Dates: First submitted 2011-01-24; First posted 2011-01-27 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Xenon; Sevoflurane; Anesthetics, Inhalation; Coronary Disease; Coronary Artery Bypass
Keywords: xenon; sevoflurane; cardiac anesthesia; CABG; Bypass surgery
MeSH Terms: conditions — Respiratory Aspiration; Coronary Disease | interventions — Xenon; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenon (Experimental): Xenon will be administered for balanced general anesthesia for CABG surgery before and after the extracorporal circulation.
  Interventions: Drug: Xenon
- Sevoflurane (Active Comparator): Sevoflurane will be administered for balanced general anesthesia for CABG surgery before and after the extracorporal circulation.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Xenon — gaseous anesthetic, dosage: 50% (v/v) in 50% oxygen, continuous application before the start and after the end of extracorporal circulation
  Arms: Xenon
Drug: Sevoflurane — inhalative anesthetic, dosage: 1.4% (v/v) in 50% oxygen/medical air , continuous application before the start and after the end of extracorporal circulation
  Arms: Sevoflurane

SUMMARY:
The aim of this study is to determine whether xenon - as compared to sevoflurane - can be applied safely in patients for general anesthesia before and after CABG implantation.

DETAILED DESCRIPTION:
The study will be conducted by two investigator types: The study enrollment and the post-anesthesia follow-up will be performed by Investigator I who is blinded to the study treatment. Investigator II will only perform general anaesthesia for CABG surgery and will therefore necessarily be unblinded to the treatment conditions.

Patients will be randomly assigned to one of the following study groups. Group 1 (Xenon) will receive xenon for maintenance of balanced anesthesia for CABG surgery before and after extracorporal circulation. Group 2 (Sevoflurane) will receive sevoflurane for maintenance of balanced anesthesia for CABG surgery before and after extracorporal circulation. During extracorporal circulation, general anesthesia will be maintained intravenously in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary artery disease scheduled for elective CABG
* Patients willing and able to complete the requirements of this study
* Ejection Fraction > 50%
* EuroSCORE ≤ 8
* men and women >= 50 yrs
* women without childbearing potential
* ASA Score II-IV

Exclusion Criteria:

* Lack of informed consent
* EuroSCORE < 8
* MMSE < 24
* Age < 50 years
* COPD GOLD > II, increased need of oxygen
* Renal dysfunction
* Liver function disorders
* Acute coronary syndrome during the last 24 hours; hemodynamic instability
* Requirement of inotropic support
* Off-pump-surgery
* Disabling neuropsychiatric disorders
* History of stroke with residuals
* Hypersensitivity to the study anaesthetics
* Increased intracranial pressure
* Pregnancy and lactation period
* Women of childbearing potential
* Presumed uncooperativeness or legal incapacity
* Participation in a concomitant trial

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety and feasibility of xenon application for general anesthesia before and after CABG implantation | an average of 4 to 6 hours
  The feasibility of xenon application compared to sevoflurane application will be assessed by:
  * The depth of anaesthesia level
  * The peri-anaesthetic respiratory profile
  * The peri-anaesthetic haemodynamic profile
  The following safety parameters will be assessed:
  * Doses and concentration of study treatments
  * Trans-esophageal echocardiography
  * Measures of renal function
  * Intra-operative blood loss and amount of transfused blood/products
  * Need for hemodynamic and inotropic support
  * The patient's regional cerebral tissue oxygenation rSO2
  * The incidence of AE and SAE

SECONDARY OUTCOMES:
Secondary efficacy and safety criteria | 6 days
  The following secondary efficacy parameters will be assessed:
  * the patients organ function status
  * The severity of postoperative critical illness
  * The incidence of Post-operative Delirium (POD)
  * The duration of postoperative intensive care unit and in-hospital stay
  Secondary safety parameters:
  * hemodynamic and respiratory profile, including vital signs
  * incidence of major adverse cardiac and cerebral events (MACCE)
  * laboratory parameters -post-operative pain
  * further AE and SAE
all cause mortality and contentment questioning | 1 year
  Patients will be contacted by telephone one year after surgery for a one year mortality and contentment examination.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Coburn, PD Dr. med., Principal Investigator — Department of Anesthesiology, University Hospital Aachen
Locations (1):
- Department of Anesthesiology, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Breuer T, Emontzpohl C, Coburn M, Benstoem C, Rossaint R, Marx G, Schalte G, Bernhagen J, Bruells CS, Goetzenich A, Stoppe C. Xenon triggers pro-inflammatory effects and suppresses the anti-inflammatory response compared to sevoflurane in patients undergoing cardiac surgery. Crit Care. 2015 Oct 15;19:365. doi: 10.1186/s13054-015-1082-7. PMID 26467531
- [Derived] Stoppe C, Fahlenkamp AV, Rex S, Veeck NC, Gozdowsky SC, Schalte G, Autschbach R, Rossaint R, Coburn M. Feasibility and safety of xenon compared with sevoflurane anaesthesia in coronary surgical patients: a randomized controlled pilot study. Br J Anaesth. 2013 Sep;111(3):406-16. doi: 10.1093/bja/aet072. Epub 2013 Apr 11. PMID 23578862